CLINICAL TRIAL: NCT04949893
Title: Causes of Chronic Pruritus: a Retrospective Study
Brief Title: Causes of Chronic Pruritus
Acronym: PRURISINE
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PRURI SINE (29BRC18.0247)
Record Dates: First submitted 2018-12-19; First posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Chronic Pruritus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to include all patients followed between 2008 and 2018 in order to analyze the etiologie of the chronic pruritus

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years old
* In patient in a day hospital or longer hospitalization in the dermatology department
* With chronic pruritus which means pruritus longer than 6 weeks without skin lesions specific to pruritic dermatitis.

Exclusion Criteria:

* Itchy dermatose
* Refusal to particpate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion of all patients with chronic pruritus followed in our dermatology department between 2008 and 2018
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
Causes of chronic pruritus | through study completion, an average of 1 year
  Analyze the etiology of chronic pruritus : uremic pruritus, cholestatic pruritus, haematologic pruritus, metabolic pruritus, neuropathic pruritus, psychogenic pruritus, idiopathic pruritus thanks to results of biological parameters, Imaging data, clinical data (for example consultation with psychiatric for psychogenic pruritus)

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France